CLINICAL TRIAL: NCT04059731
Title: Randomized, Multicentric, Double-blind, Controlled Trial of Parallel Groups to Evaluate the Non-inferiority of a Postoperative Diet With an Oligomeric-hyperprotein-normocaloric Versus Imunonutrients After Surgery for Colorectal Cancer.
Brief Title: Postoperative Diet With Hyperproteic Supplement Versus a Supplement With Imunonutrients, in Colorectal Cancer Surgery
Acronym: NUTRICOLON
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital General Universitario Reina Sofía de Murcia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NUTRICOLON
Record Dates: First submitted 2019-08-09; First posted 2019-08-16 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Nutrition Related Neoplasm/Cancer; Colorectal Cancer; Surgery--Complications; Site Infection; Nutrition Support
MeSH Terms: conditions — Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized, multicentric, double-blind, controlled with active comparator, parallel groups trial, to demonstrate non-inferiority in efficacy and therapeutic safety
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The masking procedure of the reference treatment and the study treatment will be carried out in the pharmacy service, since the packaging of the two treatments is different, brick and bottle. Pharmacy will keep the list of randomization, so at all times the pharmacy service will know which group each patient belongs to.
  Both treatments will be re-packaged in 250 ml topaz plastic bottles (Code 225433) with the same label. The re-packaging will be carried out daily in aseptic conditions and by pharmacy personnel, it will be done per patient and in no time neither the patient nor the researcher will know the group to which the patient belongs.
  In the program that the pharmacy service uses for the realization of the master formulas, the formula NUTRICOLON will be created with its corresponding procedure and label, always keeping the confidentiality of the product used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surmimed®OPD Drink (Experimental): Normocaloric oligomeric-hyperprotein supplement
  Interventions: Dietary Supplement: Nutrition supplement
- Atempero® or Impact® (Active Comparator): Inmunonutrition
  Interventions: Dietary Supplement: Nutrition supplement

INTERVENTIONS:
Dietary Supplement: Nutrition supplement — Administration twice a day of Survimed OPD or Impact/Atempero depending on arm assigned during 5 postoperative days

SUMMARY:
The study is a randomized, multicentric, double-blind, controlled with active comparator, parallel groups trial, to demonstrate the non-inferiority in efficacy and therapeutic safety of the postoperative diet with oligomeric-hyperprotéic-normocaloric supplement (group 1) versus a supplement with imunonutrients (group 2), in a multimodal rehabilitation regimen (ERAS) of colorectal surgery for colon cancer and that arrive at surgery in a normal nutritional state or without any intervention on their nutritional status, according to the scale Malnutrition Screening Tool (MST).

DETAILED DESCRIPTION:
The study is a randomized, multicentric, double-blind, controlled with active comparator, parallel groups trial, to demonstrate the non-inferiority in efficacy and therapeutic safety of the postoperative diet with oligomeric-hyperprotéic-normocaloric supplement (group 1) versus a supplement with imunonutrients (group 2), in a multimodal rehabilitation regimen (ERAS) of colorectal surgery for colon cancer and that arrive at surgery in a normal nutritional state or without any intervention on their nutritional status, according to the scale Malnutrition Screening Tool (MST). The study will be carried out in the General Surgery and Digestive Diseases Services of the following hospitals:

* Reina Sofía University General Hospital (HGURS) of Murcia.
* Sagunto Hospital, Valencia.
* University Hospital of Fuenlabrada, Madrid.

Primary objective: to demonstrate the non-inferiority in the therapeutic efficacy of a postoperative diet with an oligomeric-hyperprotéic-normocaloric supplement versus a supplement with imunonutrients, in patients under the multimodal rehabilitation regimen (fast-track) of colorectal surgery of colon cancer and who arrive at the Surgery in normal nutritional status or without any intervention on their nutritional status, according to the Malnutrition Screening Tool (MST) scale. The proportion of subjects in each research group without postoperative complications after 1 month (30 days) of surgery will be considered the main parameter of effectiveness.

Secondary Objectives: to demonstrate the non-inferiority in therapeutic safety of a postoperative diet with oligomeric-hyperprotéic-normocaloric supplement versus a supplement with imunonutrients, in a multimodal rehabilitation regimen (ERAS) of colon cancer colorectal surgery, through:

1. The evaluation in each treatment group of the oral tolerance to the supplements, considering as a total adherence if the indicated daily volume (400ml) is consumed, partial adhesion if it is half of the indicated volume (200ml) and non-adherence if it is less than 200 ml / day.
2. Comparison of the percentage of patients in each treatment group of postoperative complications according to the Clavien-Dindo classification, up to 30 days from the date of surgery.
3. Comparison of the percentage of patients in each treatment group of surgical site infection according to the classification of Centers for Disease Control and Prevention -CDC- , up to 30 days from the date of surgery.
4. The comparison in each treatment group of the percentage of patients who have required hospital readmission or have died attributed to the surgical act, up to 30 days from the date of surgery.
5. The comparison in each treatment group of the average postoperative hospital stay.
6. The evaluation in each group of treatment of analytical parameters: before nutritional supplementation prescribed by its responsible surgeon or the unit of nutrition, the day before surgery and the fifth postoperative day or the day of discharge: hemoglobin, leukocytes, lymphocytes, procalcitonin, C-reactive protein, total proteins, albumin, prealbumin, transferrin and creatinine.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years.
* Clinical diagnosis (pre-surgical) of colorectal carcinoma stage I-III, classification TNM, 6th edition.
* Normal nutritional status or without any intervention on their nutritional status, with a score lower than 2 according to the Malnutrition Screening Tool (MST) scale.
* Accepts participating in the Multimodal Rehabilitation Clinical Pathway in Patients submitted to a Bowel, Colorectal Anastomosis of HGURS.
* Accept signing informed consent.

Exclusion Criteria:

* Age under 18.
* Clinical diagnosis (pre-surgical) of colorectal carcinoma stage IV.
* ASA Staging (American Society of Anesthesiologists) IV
* Chronic renal failure in dialysis.
* Pregnant.
* Difficulty or inability to understand the purpose of the study and controls.
* Refuses to sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2019-06-20 (Actual); Primary Completion 2019-08-10 (Estimated); Study Completion 2020-06-20 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications | 30 days
  proportion of subjects in each research group without postoperative complications after 1 month (30 days) of surgery

SECONDARY OUTCOMES:
Oral Tolerance | 5 days
  The evaluation in each treatment group of the oral tolerance to the supplements, as a total adherence if the indicated daily volume (400 ml) is consumed, the partiality of half of the indicated volume (200 ml) and is not met in the minor . 200 ml / day.
Clavien-Dindo Complications | 30 days
  Comparison of the percentage of patients in each treatment group of postoperative complications according to the Clavien-Dindo classification, up to 30 days from the date of surgery.
Site Infection | 30 days
  Comparison of the percentage of patients in each treatment group of the surgical site infection according to the classification of the Centers for Disease Control and Prevention -CDC- , up to 30 days from the date of surgery
Readmission | 30 days
  The comparison in each treatment group of the percentage of patients who have required hospital readmission attributed to the surgical act, up to 30 days from the date of surgery.
Death | 30 days
  The comparison in each treatment group of the percentage of patients who have died attributed to the surgical act, up to 30 days from the date of surgery.
Hospital Stay | 30 days
  The comparison in each treatment group of the average postoperative hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Alejandro Benavides Buleje, PhD, Principal Investigator — Hospital General Universitario Reina Sofía
Locations (1):
- Hospital General Universitario Reina Sofía, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferguson M, Capra S, Bauer J, Banks M. Development of a valid and reliable malnutrition screening tool for adult acute hospital patients. Nutrition. 1999 Jun;15(6):458-64. doi: 10.1016/s0899-9007(99)00084-2. PMID 10378201
- [Background] Weimann A, Braga M, Carli F, Higashiguchi T, Hubner M, Klek S, Laviano A, Ljungqvist O, Lobo DN, Martindale R, Waitzberg DL, Bischoff SC, Singer P. ESPEN guideline: Clinical nutrition in surgery. Clin Nutr. 2017 Jun;36(3):623-650. doi: 10.1016/j.clnu.2017.02.013. Epub 2017 Mar 7. PMID 28385477
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Anderson DJ, Podgorny K, Berrios-Torres SI, Bratzler DW, Dellinger EP, Greene L, Nyquist AC, Saiman L, Yokoe DS, Maragakis LL, Kaye KS. Strategies to prevent surgical site infections in acute care hospitals: 2014 update. Infect Control Hosp Epidemiol. 2014 Jun;35(6):605-27. doi: 10.1086/676022. PMID 24799638
- [Background] Moya P, Soriano-Irigaray L, Ramirez JM, Garcea A, Blasco O, Blanco FJ, Brugiotti C, Miranda E, Arroyo A. Perioperative Standard Oral Nutrition Supplements Versus Immunonutrition in Patients Undergoing Colorectal Resection in an Enhanced Recovery (ERAS) Protocol: A Multicenter Randomized Clinical Trial (SONVI Study). Medicine (Baltimore). 2016 May;95(21):e3704. doi: 10.1097/MD.0000000000003704. PMID 27227930
- [Background] Thornblade LW, Varghese TK Jr, Shi X, Johnson EK, Bastawrous A, Billingham RP, Thirlby R, Fichera A, Flum DR. Preoperative Immunonutrition and Elective Colorectal Resection Outcomes. Dis Colon Rectum. 2017 Jan;60(1):68-75. doi: 10.1097/DCR.0000000000000740. PMID 27926559
- [Background] Wanden-Berghe C, Sanz-Valero J, Arroyo-Sebastian A, Cheikh-Moussa K, Moya-Forcen P. [Effects of a nutritional intervention in a fast-track program for a colorectal cancer surgery: systematic review]. Nutr Hosp. 2016 Jul 19;33(4):402. doi: 10.20960/nh.402. Spanish. PMID 27571677
- [Background] Calder PC. Immunonutrition in surgical and critically ill patients. Br J Nutr. 2007 Oct;98 Suppl 1:S133-9. doi: 10.1017/S0007114507832909. PMID 17922951
- [Background] Kreymann KG. Early nutrition support in critical care: a European perspective. Curr Opin Clin Nutr Metab Care. 2008 Mar;11(2):156-9. doi: 10.1097/MCO.0b013e3282f44c41. PMID 18301092
- [Background] Skipworth RJ, Fearon KC. The scientific rationale for optimizing nutritional support in cancer. Eur J Gastroenterol Hepatol. 2007 May;19(5):371-7. doi: 10.1097/MEG.0b013e3280bdbf87. PMID 17413286
- [Background] Finco C, Magnanini P, Sarzo G, Vecchiato M, Luongo B, Savastano S, Bortoliero M, Barison P, Merigliano S. Prospective randomized study on perioperative enteral immunonutrition in laparoscopic colorectal surgery. Surg Endosc. 2007 Jul;21(7):1175-9. doi: 10.1007/s00464-007-9238-4. Epub 2007 Mar 14. PMID 17356942
- [Background] Garcia-Luna PP, Parejo Campos J, Pereira Cunill JL. [Causes and impact of hyponutrition and cachexia in the oncologic patient]. Nutr Hosp. 2006 May;21 Suppl 3:10-6. Spanish. PMID 16768026
- [Background] Garcia de Lorenzo A, Alvarez Hernandez J, Planas M, Burgos R, Araujo K; multidisciplinary consensus work-team on the approach to hospital malnutrition in Spain. Multidisciplinary consensus on the approach to hospital malnutrition in Spain. Nutr Hosp. 2011 Jul-Aug;26(4):701-10. doi: 10.1590/S0212-16112011000400006. PMID 22470013